CLINICAL TRIAL: NCT01248897
Title: A Study of Biomarker Profiles in Asia Pacific erbB2+/HER2 Breast Cancer Patients Treated With Lapatinib and Other Anti-erbB2/HER2 Therapy
Brief Title: Study of Biomarker Profiles in Asia Pacific erb2+/HER2 Breast Cancer Patients Treated With Lapatinib
Acronym: BioPATH
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114021
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Neoplasms, Metastasis
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissues
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- erbB2+/Her2 Breast Cancer Patients: erbB2+/Her2 Breast Cancer Patients Treated with Lapatinib and Other Anti-erbB2/Her2 Therapy
  Interventions: Other: This study is non-interventional study, so this section is not applicable.

INTERVENTIONS:
Other: This study is non-interventional study, so this section is not applicable. — This study is non-interventional study, so this section is not applicable.

SUMMARY:
The purpose of this study is to understand how information of 3 specific biomarkers can provide guidance to physicians in the treatment of erbB2 positive breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. HER2-positive (defined as either (a) IHC3+ or (b) FISH+ in local lab) recurrent / metastatic breast cancer patients who have received treatment with lapatinib-based regimen. These are either new, current or completed cases from any of the following settings:

   * treated according to physician's clinical judgement in routine practice; or
   * treated in clinical trials with known allocation to lapatinib-based regimen; or
   * treated via lapatinib expanded access or named patient programs. These regimens should contain lapatinib as the only anti-HER2 agent.
2. Exposed to < 2 lines of trastuzumab-based regimen in the metastatic setting prior to start of lapatinib-based regimen. These regimens should contain trastuzumab as the only anti-HER2 agent.
3. Patients with an historical tumor biopsy specimen available from their primary breast cancer diagnosis. If this is not available, then at least a specimen should be available anytime during the period before the patient started on any anti-HER2 therapy.
4. Willing to give written informed consent to release the tumor biopsy specimen with corresponding clinical data. If consent could be waived according to institutional practice (eg. patient already deceased, or patient previously provided blanket consent for institution to utilize tissue/data for research purpose), this is accepted with appropriate supporting documentation.

Exclusion Criteria:

1. Patients who have been exposed to other experimental anti-HER2 therapy eg. pertuzumab, trastuzumab-DM, neratinib, ertumaxomab, AV-412, BIBW2992, CUDC-101, anti-HER2 vaccines.
2. Other primary lesions that are not of breast origin.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Asia Pacific erb2+/HER2 Breast Cancer Patients
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2010-08-17; Primary Completion 2013-12-01 (Actual); Study Completion 2014-09-05 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Time from study entry to disease progression or death from any cause, in weeks

SECONDARY OUTCOMES:
Response rate | Percentage of patients post-study entry showing complete or partial response to lapatinib
Overall survival | Time from study entry until death due to any cause, in weeks
Progression free survival | Time from first initiation of any trastuzumab-based treatment to disease progression or death from any cause, in weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Hong Kong (4):
  - GSK Investigational Site, Hong Kong
  - GSK Investigational Site, Pokfulam
  - GSK Investigational Site, Tuenmen
  - GSK Investigational Site, Wan Chai
- GSK Investigational Site, Pasay, Philippines
- GSK Investigational Site, Singapore, Singapore
- South Korea (6):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Gangwon-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Kyunggi-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Songpa-gu, Seoul